CLINICAL TRIAL: NCT02911350
Title: Phase I Study of Bi-weekly Taxol and Definitive Radiation in Androgen Ablated Locally Advanced Prostate Cancer
Brief Title: Safety Study of Combination of Hormone Therapy, Paclitaxel and Radiation Therapy to Treat Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9076
Record Dates: First submitted 2016-08-29; First posted 2016-09-22 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Paclitaxel; Albumin-Bound Paclitaxel; Radiotherapy

ARMS (1):
- Hormone Suppressors, Paclitaxel & Radiation therapy (Experimental): Hormone Suppressors: Patients may take any of the following combinations for a period of 6 months:
  1. Lupron / Flutamide
  2. Zoladex/ Flutamide
  3. Lupron/ Casodex
  4. Zoladex/ Casodex
  Paclitaxel: 30 mg/m2 twice a week administered as a one hour infusion either Monday & Wednesday or Tuesday & Thursday for eight consecutive weeks will be started within the first week of radiation therapy. Following the first 3 dose levels, the dose of Paclitaxel will be escalated to 35 mg/m2 (dose level IV), 40 mg/m2 (dose level V) & 45 mg/m2 (dose level VI).
  Radiation Therapy: 5 days a week for 8 weeks to a total dose of 66.6 to 73.8 Gray depending on when patient enter the study.
  Interventions: Drug: Hormone Suppressors; Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Hormone Suppressors
Drug: Paclitaxel
  Other Names: Abraxane
Radiation: Radiation Therapy

SUMMARY:
The purpose of this study is to determine if the combination therapy of Hormone, Paclitaxel and Radiation therapy are effective in treatment of locally advanced prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Any one or more of the following characteristics will qualify patient with T2/T3 prostate cancer for eligibility to current study:
* Biopsy proven prostate cancer with Gleason score > 7
* Pathologic staging TXN1 (on MRI or CT)
* Prostate-specific antigen (PSA) > 10 ng/ml done within a month prior to study entry (the day of first hormonal ablation) and > 10 days after prostate biopsy.

In addition patients must also have:

* Performance status < 2
* Hemoglobin > 11 grams per deciliter (g/dL), White blood cell (WBC) > 4000 and platelet count > 100.000/l
* No evidence of other synchronous primary. Prior malignancies does not exclude if the patient is disease free > 5 years.
* Prior or concurrent basal cell or non-invasive squamous carcinoma of the skin is eligible and
* Received hormone therapy with any of the following combination for less than 3 months
* Lupron / Flutamide
* Zoladex/ Flutamide
* Lupron/ Casodex
* Zoladex/ Casodex

Exclusion Criteria:

* Clinical stage T1N0, PSA < 10, and Gleason score less than 7.
* Evidence of distant metastasis
* Previous surgery for prostate cancer (radical prostatectomy).
* Current treatment with ketoconazole, cimetidine or hormone therapy for more than 3 months prior to inclusion in the protocol for prostate cancer
* Major medical or psychiatric illness, which in the investigator's opinion may prevent completion of the study and interfere with follow up.
* Bilirubin > 1.5
* Prior chemotherapy is not allowed

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2000-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) assessment | 8 weeks
  The MTD will be the lowest dose at which 2/6 or 2/3 patients experience dose limiting toxicity (DLT)
Number of participants with qualitative and quantitative toxicities | up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Sanfilippo, MD, Principal Investigator — NYU Perlmutter Cancer Center